CLINICAL TRIAL: NCT01990742
Title: Improving Palliative and End-of-Life Care in Nursing Homes
Brief Title: Improving Palliative Care Through Teamwork
Acronym: IMPACTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Helena Temkin-Greener, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PCORI-641
Record Dates: First submitted 2013-09-23; First posted 2013-11-21 (Estimated); Results first posted 2018-08-20 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-08

CONDITIONS: Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Palliative Care Team (PCTeam) (Experimental): Palliative care teams will be established and will round with residents in the intervention homes.
  Interventions: Behavioral: Palliative Care Team (PCTeam)
- Standard care (No Intervention): Usual care will be provided to residents in the control homes.

INTERVENTIONS:
Behavioral: Palliative Care Team (PCTeam) — Palliative care teams will be established and will round with residents in the intervention nursing homes.
  Arms: Palliative Care Team (PCTeam)

SUMMARY:
One in three Americans dies in a nursing home (NH) or in a hospital, shortly following transfer from a long-term care facility. The proportion of deaths occurring in NHs is projected to increase to 40% by 2020. Excellence in palliative and end-of-life (EOL) care must become a priority for these long-term care institutions. However, findings from NHs point to high incidence of pain and poor management of other symptoms and excessive reliance on hospitalizations, indicating inadequate EOL care quality. Expert opinion and research have suggested that poor EOL quality in NHs may be due to lack of palliative care training among staff and absence of EOL care protocols or guidelines, but research demonstrating that attention to these factors improves outcomes is absent. While dedicated care teams have been shown to improve outcomes for NH residents in need of specialized care, the impact of palliative care teams in improving resident outcomes has remained largely unstudied and untested. This will be the first randomized controlled trial to evaluate the impact of palliative care teams (PCTeam) on resident and staff outcomes, and care processes, in NHs.

Our objective is to demonstrate, using a randomized controlled trial design and a difference in difference analytic approach, that nursing home-based palliative care practice guidelines implemented through PCTeams will improve quality of care processes and outcomes for residents at the end of life.

We will adapt existing palliative care guidelines for EOL care, endorsed by the National Quality Forum (NQF), to the NH environment, deploy the adapted practice guidelines through a PCTeam model, and evaluate the effectiveness of this intervention on resident EOL outcomes and staff care processes and outcomes. The specific aims (SA) will address the following questions:

SA 1: Is PCTeam intervention effective in improving NH residents' EOL outcomes?

SA 2: Is PCTeam intervention effective in improving NH staff EOL care processes and outcomes?

In the context of these specific aims we will test the following hypotheses:

H1: Residents in NHs in the intervention arm, compared to the control, will achieve better EOL risk-adjusted outcomes and care processes with regard to:

* Pain
* Dyspnea
* Depression
* In-hospital deaths
* Hospitalizations
* Advance directives

H2: Direct care staff in NHs in the intervention arm, compared to the control, will achieve better EOL processes and outcomes measured by:

* Assessment of EOL symptoms
* Delivery of EOL care
* Communication/coordination among providers
* Communication with residents/families
* Teamwork effectiveness
* Staff satisfaction

H3: Family caregivers of decedent residents in the intervention NHs, compared to the control, will report receiving more patient and family centered care as measured by higher levels of satisfaction with:

* Shared decision making between providers, the patient and the family
* Care that is respectful of the patient wishes and dignity
* Attention to the emotional and spiritual needs of the family.

  31 NHs in upstate New York have been recruited for the study (letters of support). Stakeholders include residents, family members, staff, policy makers, and others. The intervention will deploy theTeamSTEPPS, a team development model created by the Department of Defense and the Agency for Healthcare Research and Quality.

ELIGIBILITY:
Inclusion Criteria:

* long-stay nursing home residents (>90 days)

Exclusion Criteria:

* rehabilitative, post-acute residents (<90 days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-09-27 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helena Temkin-Greener, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester School of Medicine and Dentistry, Rochester, New York, United States

REFERENCES:
- [Derived] Ryan RE, Connolly M, Bradford NK, Henderson S, Herbert A, Schonfeld L, Young J, Bothroyd JI, Henderson A. Interventions for interpersonal communication about end of life care between health practitioners and affected people. Cochrane Database Syst Rev. 2022 Jul 8;7(7):CD013116. doi: 10.1002/14651858.CD013116.pub2. PMID 35802350

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Nursing Homes, not individual participants, were enrolled in this RCT study, and were the unit of intervention. However, the outcomes analysis was performed on decedents who were cared for in the enrolled Nursing Homes.
Units Other Than Participants: Nursing Homes
Groups:
- Palliative Care Team (PCTeam): Palliative Care Team (PCTeam): Palliative care teams will be established and will work with residents in the intervention nursing homes.
Period: Overall Study
Arm/Group | Palliative Care Team (PCTeam) | Standard Care
Started | 3259; 16 Nursing Homes (This is a facility-level intervention, access to individual level records occurred via MDS data only) | 4331; 15 Nursing Homes (This is a facility-level control , access to individual participants occurred only via MDS records.)
Completed | 2852; 14 Nursing Homes (Fourteen facilities completed the intervention.) | 2978; 11 Nursing Homes (Eleven nursing homes completed the control group /usual care allocation.)
Not Completed | 407; 2 Nursing Homes | 1353; 4 Nursing Homes
Not completed — Withdrawal by facility | 407 | 1083
Not completed — Facility closed | 0 | 270

BASELINE CHARACTERISTICS:
Population: All decedents with data who resided in assigned facilities.
Groups:
- Total: Total of all reporting groups
Arm/Group | Palliative Care Team (PCTeam) | Standard Care | Total
Number analyzed (Participants) | 2852 | 2978 | 5830
Age, Continuous [Mean (Standard Deviation); unit: years] | 86.0 (8.9) | 86.2 (9.0) | 86.1 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Individual participants were not enrolled; we report here the gender of the nursing home residents who died during the study period in our enrolled facilities, as recorded in the MDS data set used for the outcomes analyses.
  Participants
    Female | 1813 | 1930 | 3743
    Male | 1039 | 1048 | 2087
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Individual participants were not enrolled; we report here the ethnicity of the nursing home residents who died during the study period in our enrolled facilities, as recorded in the MDS data set used for the outcomes analyses.
  Participants
    Hispanic or Latino | 1 | 18 | 19
    Not Hispanic or Latino | 2851 | 2960 | 5811
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Individual participants were not enrolled; we report here the racial distribution of the nursing home residents who died during the study period in our enrolled facilities, as recorded in the MDS data set used for the outcomes analyses.
  Participants
    American Indian or Alaska Native | 22 | 22 | 44
    Asian | 11 | 11 | 22
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 108 | 153 | 261
    White | 2711 | 2792 | 5503
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — The nursing home in which each decedent received care serves as the geographic location for this baseline measure.
  participants
    United States | 2852 | 2978 | 5830

OUTCOME MEASURES:

1. Primary Outcome: Hospital Site of Death: Number of Decedents Cared for in an Enrolled and Assigned NH Facility, Who Were Transferred to a Hospital and Died in the Hospital During the Study Period
Description: This outcome measure, Hospital Site of Death, assesses whether death occured in a nursing home or in a hospital following transfer from the nursing home, among nursing home residents who were cared for in an enrolled facility.
Time Frame: 1 year
Population: Nursing home residents cared for in an assigned facility, who died during the study timeframe
Measure: Count of Participants; unit: Participants
Arm/Group | Palliative Care Team (PCTeam) | Standard Care
Number analyzed (Participants) | 2852 | 2978
Participants | 579 | 441
Statistical Analysis 1: Comparison: Palliative Care Team (PCTeam) vs Standard Care; Test type: Other; p > 0.05, MOnte carlo simulation

2. Secondary Outcome: Hospitalizations
Description: Number of hospitalizations in the last 90 days of life among decedents being cared for in the enrolled nursing homes
Time Frame: The last 90 days of life
Population: Decedents with data on hospitalizations in the last 90 days of life
Measure: Mean (Standard Deviation); unit: Mean number of hospitalizations
Arm/Group | Palliative Care Team (PCTeam) | Standard Care
Number analyzed (Participants) | 1907 | 1930
Mean number of hospitalizations | 0.34 (0.69) | 0.29 (0.62)
Statistical Analysis 1: Comparison: Palliative Care Team (PCTeam) vs Standard Care; Test type: Other; p > 0.05, Monte carlo simulation

3. Other Pre Specified Outcome: Number of Nursing Home Residents in Moderate-to-severe Pain
Description: Presence of moderate-to-severe pain within 6 months of the date of death, among decedents cared for in the enrolled nursing homes. The verbal descriptor pain scale, where the resident is asked to rate the intensity of their worst pain in the last five day was most often used, where 0 = no pain, 1 = mild pain , 2 = moderate pain, 3 = severe pain, 4 = very severe pain, and 9 = unable to answer. Lower numbers (0 or 1 ) on the scale are preferred, and a lower percentage of residents reporting pain intensity in the moderate or higher ranges is a better outcome. The verbal descriptor scale can be shared with elders verbally, as the name implies, or by asking the resident to point to a setting on a visual thermometer with these word choices.
Time Frame: up to 6 months prior to death
Population: Decedents cared for in assigned nursing home facilities for whom data on pain was available
Measure: Count of Participants; unit: Participants
Arm/Group | Palliative Care Team (PCTeam) | Standard Care
Number analyzed (Participants) | 1844 | 1851
Participants | 235 | 218
Statistical Analysis 1: Comparison: Palliative Care Team (PCTeam) vs Standard Care; Test type: Other; p > 0.05, Monte carlo simulation

ADVERSE EVENTS:
Time Frame: 1 year
Description: We only collected and used data on decedents in our enrolled nursing homes, therefore ALL individual level outcomes measures are based on residents who died during the study period. However, the intervention was not at the individual level, but rather a facility-level. The study was not directly associated with, or a cause of, any of these deaths. Rather, we aimed to teach nursing home staff in the intervention facilities how to improve the quality of care for residents who were dying.
Arm/Group | Palliative Care Team (PCTeam) | Standard Care
All-Cause Mortality (participants affected / at risk) | 2852/2852 | 2978/2978
Serious Adverse Events (participants affected / at risk) | 2852/2852 | 2978/2978
Other Adverse Events (participants affected / at risk) | 0/2852 | 0/2978
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palliative Care Team (PCTeam) (N=2852) | Standard Care (N=2978)
Death from causes not associated with the study (General disorders) | 2852 (2852) | 2978 (2978) — We based our comparative outcomes assessment using the MDS 3.0 data available only from decedents cared for by the enrolled nursing homes. Therefore, all individual-level data was obtained from patients who suffered death, within the study timeframe.

LIMITATIONS AND CAVEATS:
1. We were unable to distinguish the relative importance of the individual intervention components.
2. Our findings were confined to regional facilities, and may not be generalized elsewhere.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No